CLINICAL TRIAL: NCT04029701
Title: Clinical Observation on the Treatment of Motor and Sensory Dysfunction After Stroke With Ruyizhenbao Pill
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-K-38
Record Dates: First submitted 2019-07-07; First posted 2019-07-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Post-stroke Patients With Motor and Sensory Dysfunction
Keywords: Ruyizhenbao Pill; Post-stroke; Motor dysfunction; Sensory dysfunction
MeSH Terms: conditions — Neurologic Manifestations | interventions — Research Design; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This Trials is a randomly controlled, double-blinded and placebo-controlled trial.And the methodology team of Guangdong Provincial Hospital of Chinese Medicine is responsible for the editing of blindness.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research group (Experimental): Subjects who are recruited into this group are asked to take the Ruyizhenbao Pill on the basis of routine internal medicine and rehabilitation treatment.
  P.S. Ruyizhenbao Pills are provided by Jinhe Tibetan Pharmaceutical Co., Ltd. Chinese national medicine permission number:Z63020289、Z63020064. Medication method: oral 4 pills once, twice a day, 4 weeks in a row.
  Interventions: Drug: Ruyizhenbao Pill
- Control group (Placebo Comparator): Subjects who are recruited into this group are asked to take the placebo of Ruyizhenbao Pill on the basis of routine internal medicine and rehabilitation treatment.
  P.S. Placebo is provided by Jinhe Tibetan Pharmaceutical Co., Ltd.，which is made of malt dextrin as a matrix, similar shape and same color to the Ruyizhenbao Pill. Medication method: oral 4 pills once, twice a day, 4 weeks in a row.
  Interventions: Drug: Placebo of Ruyizhenbao Pill

INTERVENTIONS:
Drug: Ruyizhenbao Pill — Ruyizhenbao Pills are provided by Jinhe Tibetan Pharmaceutical Co., Ltd. Chinese national medicine permission number:Z63020289、Z63020064. Medication method: oral 4 pills once, twice a day, 4 weeks in a row.
  Other Names: Research group
  Arms: Research group
Drug: Placebo of Ruyizhenbao Pill — Placebo is provided by Jinhe Tibetan Pharmaceutical Co., Ltd.，which is made of malt dextrin as a matrix, similar shape and same color to the Ruyizhenbao Pill. Medication method: oral 4 pills once, twice a day, 4 weeks in a row.
  Other Names: Control group
  Arms: Control group

SUMMARY:
Many years of clinical practice experience has found that Ruyi treasure pill can be used to treat nerve meridian injury caused by cerebrovascular disease, but in the end, the clinical efficacy is still lacking systematic clinical evidence-based medical research data. Based on this, the clinical observation of Ruyi treasure pill in the treatment of post-stroke motor and sensory dysfunction was carried out to verify its clinical location, to provide evidence for the application of clinical subdivision of later products and two development of products, and to publish academic papers on the expected research results.

ELIGIBILITY:
Inclusion Criteria:

1. Compliance with stroke diagnostic criteria;
2. The course of the disease is 15 days to 6 months;
3. People who are conscious and have no severe cognitive impairment, and those who cooperate with examination and treatment;
4. Age 20 to 80 years old;
5. Sign an informed consent and participate voluntarily in the study.

Exclusion Criteria:

1. Diseases such as brain tumours, traumatic brain injury, brain parasitic diseases and metabolic disorders have been confirmed by examination;
2. Combining patients with severe heart, liver, kidney, hematopoietic and endocrine systems, gastrointestinal diseases, etc.;
3. Those who are not aware or concoced due to more severe cognitive impairment and complete aphasia;
4. People who are allergic to the drug or are allergic to multiple medications.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor function change | The simplified Fugl-Meyer motion function scale will be tested totally twice,separately at before taking drugs, 4 weeks and 8 weeks after taking drugs so as to compare changes among three time points.
  Using Simplified Fugl-Meyer motion function assessment method to assess the motor function of affected side.The total score of Fugl-Meyer motor function assessment scale is 100 points，50 items intotal with 2 points each. Accordding to the quality of mission completion，evaluater mark score of "0","1",2".Among them, 33 items are evaluated for upper limbs, with a total score of 66 points. And 17 items are evaluated for lower limbs,with a total score of 34 points.The higher the scores, the better motor function.If the total score is less than 50, it means severe dyskinesia.If the total score is between 50-84, it means obvious movement disorder.If the total score is between 85-95, it means moderate dyskinesia.If the total score is between 96-100, it means mild dyskinesia.
Sensory function change | Simplified Fugl-Meyer sensory function scale will be tested before taking drugs, 4 weeks and 8weeks after taking drugs so as to compare changes at three time points.Three times in total.
  Using Simplified Fugl-Meyer sensory function assessment scale to assess the sensory function of affected side,which includes light touch and proprioception. Light touch includes 4 parts, which are respectively upper arm, palm, thigh, foot. Proprioception includes 7 parts,which are respectively shoulder, elbow, wrist, thumb, knee, ankle, toe joint. The total score of each part is 2,the total scores of this scale is 22."0" score means no feeling，"1" score means feeling allergic or diminished，"2"scores means normal feeling.The sum of the scores of each part is the total score. The higher the total scores,the better the sensory function.
Activity of daily living(ADL)change | Modified Barthel Index will be tested before taking drugs, 4 weeks and 8weeks after taking drugs.Three times in total.
  Using Modified Barthel Index to assess the activity of daily living. TheMBI scale includes 11 items with total scores of 100. Evaluation is based on the actual situation of the patient.The sum of the scores of each item is the total score,and the lowest score is"0",the highest scores is"100".If the scores is between 0-20 points,it means extremely severe dysfunction.If the scores is between 25-45 points,it means severe dysfunction.If the scores is between 50-70 points it means moderate functional defects.If the scores is between 75-95 points,it means mild functional defects.If the scores is 100 points,it means ADL self-care.The higher the total scores,the better the ADL.
Survival Quality Score change | Special scale of quality of life will be tested before taking drugs, 4 weeks and 8weeks after taking drugs so as to compare changes at three time points.Three times in total.
  Special scale of quality of life is used to test the survival quality this week. 3 selected questions are evalusted and there are 5 selections for each question. "1" means "Exactly"，"2" means "Basically"，"3"means "Not sure"，"4"means "Basically not"，"5"means "Absolutely not".The sum of the scores of each question is the total score. The higher the total scores,the better the survival quality.
Berg Balance Function change | Berg Balance Function Scale will be tested before taking drugs, 4 weeks and 8weeks after taking drugs so as to compare changes at three time points.Three times in total.
  Berg balance function scale is to assess the balance function.It contains 14 instructions with total scores of 56.Each instruction includes 5 selections respectively for"0","1","2","3","4".The sum of the scores of each instruction is the total score. The higher the total scores,the better the balance function.
Painful degree change | VAS will be tested before taking drugs, 4 weeks and 8weeks after taking drugs so as to compare changes at three time points.Three times in total.
  Visual analog scale(VAS) is used to test the painful degree. It contains 0-10 scores,while "0"means no pain, "10"means most severe painful.The higher the scores,the more painful.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ling SS, Pan RH, Zhan LC, Li M, Yang ZJ, Yang HD, Chen HX. Ruyi Zhenbao Pills for Patients with Motor and Sensory Dysfunction after Stroke: A Double-Blinded, Randomized Placebo-Controlled Clinical Trial. Chin J Integr Med. 2022 Oct;28(10):872-878. doi: 10.1007/s11655-022-3577-9. Epub 2022 Jun 20. PMID 35723814